CLINICAL TRIAL: NCT02553187
Title: A Prospective, Randomized, Controlled, Multicenter Study of Kanglaite Injection for the Treatment of Cancer Cachexia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Kanglaite Pharmaceutical Co.Ltd (Other)
Collaborators: H & J CRO International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KLT201401
Record Dates: First submitted 2015-09-09; First posted 2015-09-17 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Cancer Cachexia
MeSH Terms: interventions — kang-lai-te

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment group (Experimental): Kanglaite Injection plus standard therapy.
  Interventions: Drug: Kanglaite Injection
- Control group (No Intervention): Blank control and standard therapy.

INTERVENTIONS:
Drug: Kanglaite Injection — 200 mL, slow IV drip, once daily for 14 consecutive days, subsequent courses repeated after a 7-day interval.
  Subjects will be treated for 4 courses (12 weeks).
  Other Names: Coicis Oil injection
  Arms: Treatment group

SUMMARY:
The purpose of the study is to explore the efficacy and safety of Kanglaite Injection in the treatment of patients with late-stage cancer cachexia.

DETAILED DESCRIPTION:
The study is a multicenter, prospective, randomized controlled study. The planned sample size is 160 subjects. These subjects will be randomized (1:1) to treatment group (i.e., standard therapy plus Kanglaite Injection) or control group (i.e., standard therapy plus blank control). The study population includes the patients with non small cell lung cancer (adenocarcinoma), colorectal carcinoma and pancreatic carcinoma, who are complicated with cachexia.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed patients with stage III-IV non-small cell lung cancer (adenocarcinoma), colorectal carcinoma or pancreatic carcinoma, who are not eligible for surgery, interventional treatment and radiation therapy;
2. Confirmed patients with cachexia: weight loss greater than 5% in last six months, or BMI<20kg/m2 and weight loss greater than 2%, or in accordance with the diagnosis of sarcopenia and weight loss greater than 2%;
3. Patients who are not being treated with chemotherapy should have completed chemotherapy 14 days before randomization of this study;
4. For patients who are being treated with chemotherapy, the chemotherapy regimen should be confined to the regimens specified in the protocol; and the chemotherapy regimen, in general, are not allowed to be changed during the study period;
5. Patients are conscious and able to cooperate with the doctor to complete the disease-related examinations and evaluations;
6. ECOG performance status (PS) 0-3 for those who are not treated with chemotherapy; and ECOG PS 0-2 for those who are being treated with chemotherapy;
7. Expected survival period is more than 4 months;
8. Male or female aged 18 - 75 years;
9. Patients who are willing to participate in the study and sign the informed consent form.

Exclusion Criteria:

1. Any pathological type of non-small cell lung cancer (NSCLC) except adenocarcinoma;
2. Patients who are being treated with chemotherapy, the chemotherapy regimen is not among the regimens specified in the protocol;
3. Patients with cachexia caused by other reasons, e.g. severe hepatic dysfunction [Aspartate transaminase(AST)/Cerealthirdtransaminase(ALT) >5 times the ULN], severe renal dysfunction (Cr >1.5 times the ULN), uncontrolled thyroid disease, New York Heart Association (NYHA) class III-IV heart failure, AIDS etc.;
4. Any condition that may hinder the subject's completion of the study, including but not limited to severe uncontrollable organic diseases or infection, unstable angina pectoris, congestive heart failure, etc.;
5. Patients who are being treated with other anticancer traditional Chinese medicine (TCM), or those who may be treated with TCM after enrollment;
6. Patients with severe hepatic dysfunction: Scr >=1.5 times the ULN, ALT/AST/alkaline phosphatase (ALP) >=5 times the ULN, total bilirubin (TBIL) >=1.5 times the ULN;
7. Patients with severe abnormal lipid metabolism [TC>300mg/dl or Triglyceride(TG) >2.5 times the ULN], or those who are in lipid-lowering therapy;
8. Known or suspected diagnosis of metastatic encephaloma;
9. In treatment of or plan to receive treatment of molecular targeted drugs, eg,epidermal growth factor receptor

   - tyrosine kinase inhibitor (EGFR-TKI), anaplastic lymphoma kinase (ALK) inhibitor, anti-angiogenic agents (including monoclonal antibodies and endostatin), and cetuximab;
10. Patients present with an ECOG score>2 and require treatment of chemotherapy;
11. Patients with allergies or intolerability to the investigational product or its excipients;
12. Patients who are currently included in other clinical trials on antineoplastic drugs;
13. Patients who are not able to provide the Informed Consent Form (ICF);
14. Expected survival period is less than 4 months;
15. Female patient is pregnant or breast-feeding, and those patients at childbearing age who are not willing to use methods of contraception (including males);
16. Patients with symptomatic, uncontrolled nervous disorders, mental illness or psychiatric disorder;
17. Any condition, in the investigator's opinion, is not in the best interest of the subject (e.g., harming the subject's health) or potentially interferes with the evaluation of treatment according to this protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2017-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Body weight | 77days
Lean body mass | 77days

SECONDARY OUTCOMES:
Progression-free survival rate (PFS) | 77days
Eastern Cooperative Oncology Group score (ECOG) | 77days
Quality of life score (QOL) | 77days
Survival curve | 77days
Overall Survival (OS) | 77days
Body Mass Index (BMI) | 77days
Serum albumin | 77days
Serum Prealbumin | 77days
Serum Lactic Acid | 77days
Incidence of myelosuppression (%) | 77days

CONTACTS AND LOCATIONS:
Overall Officials: Shiying YU, Principal Investigator — Tongji Hospital
Locations (1):
- Cancer Center, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China